CLINICAL TRIAL: NCT01584271
Title: Phase II 3 Arm Double Blinded Clinical Study Evaluating the Pain Killing and Healing Time of Botanical Ear Drops, Ear Comfort(TM), in Severe External Ear Infection (AOE) Patients, Compared to Dex-Otic(R) and Otidin(R)
Brief Title: Study of Ear Comfort Ear Drops to Treat AOE Cases Compared to DexOtic & Otidin(R)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011058
Record Dates: First submitted 2012-04-05; First posted 2012-04-24 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2012-04

CONDITIONS: Acute Otitis Externa
Keywords: AOE; Ear Comfort; Dex Otic; Otidin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 Dex-Otic ear drops (Active Comparator): Dex-Otic(R) ear drops are used for pain relief and treating ears of AOE patients. It contains: Dexamethasone Sodium Phosphate 1 mg; Neomycin sulfate 5 mg; Polymyxin B sulfate 10,000 units. It
  Interventions: Device: Natural Ear Comfort(TM), a botanical ear drops product
- 3 Ear Comfort(TM) ear drops (Experimental): Natural Ear comfort(TM) ear drops contains Chamomile extract and Thyme oil in anhydrous glycerin for pain relief and ear healing.
  Interventions: Device: Natural Ear Comfort(TM), a botanical ear drops product
- 1 Otidin(R) ear drops (Active Comparator): Otidin(R): Ear drops containing Tetracaine HCL 0.5%; antipyrine 5% in anhydrous glycerin for pain relief in AOE patients.
  Interventions: Device: Natural Ear Comfort(TM), a botanical ear drops product

INTERVENTIONS:
Device: Natural Ear Comfort(TM), a botanical ear drops product — Ear Comfort(TM): active ingredients - Thyme essential oil & Camomile extract. Inactive ingredients: anhydrous glycerin and a small quantity of surfactant.
  Dex-Otic(R): Dexamethasone sodium phosphate 1mg; neomycin sulfate 5mg; polymixin B sulfate 10,000 units.
  Inactive ingredients: propylene glycol, sodium acetate anhydrous, phenyl mercuric acetate, purified water.
  Otidin(R): Tetracaine HCL 0.5%; antipyrine 5% in anhydrous glycerin.
  Other Names: 1 local pain killer; 2 antibiotics & steroid anti-inflamatory ear drops; 3 Ear Comfort(TM) botanical ear drops

SUMMARY:
Phase II 3 arm double blinded clinical study, to evaluate pain killing and healing time of Botanical Ear Drops, Ear Comfort™, in Severe External Ear Infection (AOE) patients in comparison to Dex-Otic® and Otidin®.

Study Outcome (hypothesis): if Ear Comfort™ proves to perform as well as Dex-Otic, then ENT's and family doctors will have a botanical non-antibiotic product that does not promote the formation of antibiotic-resistant infections and may be given to anti-biotics sensitive patients.

Ear comfort™ is pharmacologically stable for at least 3 years on the shelves.

DETAILED DESCRIPTION:
Severe External Ear Infection (AOE) also known as Swimmer's ear, is an abundant microbiological contamination disease of the outer ear canal. It causes severe pains and accumulation of fluids in the ear. In some cases it may compromise the hearing. Swimming in contaminated water or cleaning the ear with a hard subject are only two examples of what may cause AOE. The main Pathogenes causing the disease are Gram negative of which Pseudomonas aeruginosa is the most abundant. Occasionally it is a fungoid contamination with Aspergillus Niger being the most abundant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AOE.
* AOE patient determined by ear canal obstruction, exudates and pain.
* Males and Females between 18 and 65 years of age.
* Patients willing to refrain from using any ear drops products for the entire duration of the study. - - Subjects are willing to use the full 4 steps protocol
* Written informed consent has been obtained.

Exclusion Criteria:

* Known allergy or sensitivity to Chamomile extract or essential oils.
* Injury to tympanic membrane.
* Medical or psychiatric conditions that affect the patient's ability to give informed consent, or complete the study.
* Pregnant or lactating females.
* Use of ear drops or antibiotic or analgesic medications within the last 4 weeks prior to enrolment to the study.
* Other known diseases, including severe allergy, chronic liver or kidney disease, malignancy or contagious diseases, such as HIV or hepatitis.
* Alcohol or drug abuse, according to assessment by the investigator.
* Participation in other clinical trial within the last 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Ear Comfort(TM) kills pain in AOE patients within how many hours? | 12 months
  Comparing Ear Comfort(TM) botanical ear drops performance in killing pain in AOE patients to Dex-Otic and Otidin Will be measured by Pain Scores on the Visual Analog Scale. The patients will score their pains on a patient's diary document. A professional medical statitician expert will make the anlysis.

SECONDARY OUTCOMES:
Does Ear Comfort(TM) heal the inflamation in AOE patients? | 12 months
  Performance of Ear Comfort(TM) ear drops, Dex-Otic and Otidin in healing AOE patients ear will be measured by: - reducing microbiological load, patient's compliance and ENT expert/s check of the year during the treatment period and 7 days after stopping the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Guttman, MD, Principal Investigator — Maccabi Healthcare Services, Israel
Locations (1):
- "Maccabi" Clinic, Gedera, Israel